CLINICAL TRIAL: NCT01826942
Title: Scar Prevention Using Fractional Carbon Dioxide Laser Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Cooperation stooped with PI
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-ABU-UP-13-01
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Scar Prevention
Keywords: Scar prevention; CO2 fractional laser

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thin skin (Experimental): Single fractional CO2 treatment at surgical area closure procedure on thin skin
  Interventions: Device: Lumenis UltraPulse single fractional CO2 laser treatment thin skin
- Thick skin (Experimental): Single fractional CO2 treatment at surgical area closure procedure on thick skin
  Interventions: Device: Single fractional CO2 treatment at surgical area closure procedure on thick skin

INTERVENTIONS:
Device: Lumenis UltraPulse single fractional CO2 laser treatment thin skin
  Arms: Thin skin
Device: Single fractional CO2 treatment at surgical area closure procedure on thick skin
  Arms: Thick skin

SUMMARY:
In this study the investigators intend to determine the impact of fractional CO2 laser treatment on the edges of a fresh wound during surgical area closure on thin skin (e.g. face, hands, arms, thorax, etc.) and on thick skin (abdominoplasty procedure) on scar formation. The investigators will also evaluate the effect of shallow fractional laser treatment versus deep parameters settings. If effective treatments could be performed at time of surgery, this would result in both time and cost saving to the patient and to the healthcare system and will improve patient's self-image post surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Male or Females
* At least 18 and no more than 65 years old
* The surgical area closure in these subjects should be at least 4cm
* Type of surgery scheduled:

Site 1: Surgical area closure on thin skin, including areas that require motion (e.g. face, hands, arms, thorax, etc.) Site 2: Surgical area closure on thick skin (abdominoplasty procedure)

* Willing to comply with study dosing and complete the entire course of the study

Exclusion Criteria:

* Active bacterial, fungal, or viral infection in the treatment area
* Active cold sores, or herpes in the treatment area
* Recent excessive exposure to sunlight or artificial UV light (e.g.: use of tanning beds/booths and/or sunbathing) or expectations of tanning during the time of the study
* History of skin cancer, unless the surgical procedure of issue is for cancer treatment purposes.
* History of or the presence of any skin condition/disease that might interfere with the diagnosis or evaluation of study parameters (i.e., atopic dermatitis, eczema, psoriasis)
* Treatment with a systemic retinoid within the past year (e.g., Accutane®, Roche Dermatologics)
* History or presenting with a keloid scar
* Any current or recent treatment for cancer, unless the surgical procedure of issue is for cancer treatment purposes.
* Any uncontrolled systemic disease. A potential subject in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study
* Significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
* Subject planning any other cosmetic procedure to the study area during the study period, other than the treatments that will be performed by the investigator
* Female subject who is pregnant, nursing an infant or is less than 6 months after termination of breast feeding
* Small surgical closure (<4cm)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Scar appearance by blinded evaluation of photographs of the three month follow-up visit | three month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Ronald L. Moy, M.D., Beverly Hills, California, United States